CLINICAL TRIAL: NCT01295775
Title: A Multicentre, Double-Blind, Randomised, Placebo Controlled Study of the Activity of Sulodexide in Diabetic Patients With Mild to Moderate Non-Proliferative Retinopathy
Brief Title: Diabetic Retinopathy Sulodexide Study
Acronym: DRESS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Ji Hun Song, Assistant professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DRESS_Korea
Record Dates: First submitted 2010-07-22; First posted 2011-02-15 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2012-11

CONDITIONS: Diabetic Retinopathy
Keywords: diabetic retinopathy; sulodexide; hard exudates; microaneurysms; hemorrhages; intraretinal microvascular abnormalities
MeSH Terms: conditions — Diabetic Retinopathy; Microaneurysm; Hemorrhage | interventions — glucuronyl glucosamine glycan sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sulodexide group (Active Comparator): 50 mg of sulodexide a day will be administered by oral route (1+1 capsule/day) for 360 days
  Interventions: Drug: sulodexide
- Placebo group (Placebo Comparator): Sulodexide placebo will be administered at the same schedule (1+1 capsule/day) and for the same lengths of time (for 360 days) as Sulodexide group
  Interventions: Drug: sulodexide

INTERVENTIONS:
Drug: sulodexide — A (SULODEXIDE GROUP):
  50 mg a day by oral route (1+1 capsules/day) for 360 days
  B (PLACEBO GROUP):
  Sulodexide placebo at the same schedule dosage and for the same lengths of time as group A.
  Other Names: vessel due F

SUMMARY:
The aim of this phase 2 controlled placebo study is to assess the effectiveness of Sulodexide in the treatment of non proliferative (background) retinopathy in patients with Type 1 and Type 2 Diabetes Mellitus.

This is a multicentre, double-blind, randomised study involving patients affected by non proliferative (background) diabetic mild to moderate retinopathy.

This study will involve 130 patients (65 for each group). At baseline visit (T0), the Investigator will grade the ocular lesions due to diabetic retinopathy according to color fundus photographs and the fluorescein angiography examination. He will subsequently send the negatives of photographs and the images -or negatives when available- of fluorescein angiography to an off-site Assessor -unaware of the Investigator assessment- nominated to confirm the quality of the images and the grade of the lesions. After positive assessment of the Investigator, at T0 the eligible patient will be blindly allocated to one of the 2 treatment groups according to a computer-generated randomisation list provided by the Sponsor.

The following treatments will be administered for 360 days:

A (SULODEXIDE GROUP): 50 mg a day by oral route;

B (PLACEBO GROUP): Sulodexide placebo at the same schedule and for the same lengths of time as group A.

Before breaking the randomisation code at the end of the study, an independent off site assessor will evaluate the photographs according to the Airlie House Classification and following modification by Early treatment Diabetic Retinopathy Study (ETDRS) and fluorescein angiography according to ETDRS.

DETAILED DESCRIPTION:
Diabetic retinopathy is the leading cause of blindness in adults (20 to 74 years old) in the industrialised countries, affecting from 2 to 5% of entire population. All the complications of diabetes such as diabetic retinopathy, are caused by the chronic hyperglycaemia. Although a good metabolic control with therapy lowers the blood glucose levels enough to preserve life, this does not permit complete euglycemia nor prevent the long-term complications of chronic supernormal levels of blood glucose. The excess glucose causes flux through the polyol pathway, which results in structural tissue modifications.

Diabetic retinopathy is mainly a vascular disease, primarily affecting the capillaries. The first ultrastructural and microscopic changes reported are retinal capillary basement membrane thickening and pericyte degeneration, both of which compromise the integrity of the capillary wall, followed by pericyte loss.

The glycosaminoglycans (GAGs) of the basal membrane are progressively substituted by collagen, leading to a modification in vascular permeability due to the altered anionic charge. These changes lead to the clinical appearance of vascular leakage from retinal capillaries followed by microaneurysms. The lack of integrity of the vessel wall leads to haemorrhages, and to microthrombosis, which are responsible for the first ischemic lesions. If the vascular leakage lasts for a long time, the lipidic fraction of leaked plasma deposits in the retina forming hard exudates.

The substitution of GAGs by collagen leads to a basal membrane thickening also in the kidney. As in the retina, the modification of permeability occurs in the renal glomeruli and induces the selective loss of proteins (albuminuria).

Recent papers show a specific modification in GAGs metabolism occurring in diabetic patients that could be the common pathogenetic mechanism of vascular diabetic failure. Therefore, diabetic retinopathy and diabetic nephropathy may be regarded as the result of the alteration of a common underlying molecular mechanism whose expression is the depletion of GAGs from the basement membrane in both retinal and glomerular capillaries. In agreement with the previous statement, the Wisconsin Epidemiologic Study of Diabetic Retinopathy concluded that microalbuminuria is associated cross-sectionally with the presence of retinopathy in diabetic patients.

The progress of the clinical symptoms of the disease despite glycaemic therapy points to address the research towards new drugs able to slow or reverse the vessel micro-abnormalities responsible for the microangiopathy typical of diabetic retinopathy. Furthermore, the similarities of the vessel lesions between diabetic retinopathy and diabetic nephropathy suggest that new molecules effective in one of the two conditions should be effective in the other pathology as well.

Sulodexide (fast moving heparin fraction 80% and dermatan sulfate 20%) is a GAG with a high trophism for vessel wall. Clinical studies showed its efficacy in decreasing both microalbuminuria and macroalbuminuria in diabetic patients, suggesting that it could be able to slowdown the nephropathy progression, actually by partially restoring the glomerular GAGs content.

Preliminary observations regarding the use of Sulodexide in patients suffering from diabetic retinopathy show significant reduction in hard exudates, thus indirectly pointing out a benefit of this GAG at the retinal capillary level.

Based on the above mentioned physiopathological considerations and experimental findings, the investigators deem appropriate to evaluate the effects of Sulodexide on the diabetic retinopathy by the present multicentre, double-blind, placebo-controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 1 or Type 2 Diabetes Mellitus
* Diabetes under good control with drugs for at least 6 months (Glycosylated hemoglobin <9% )
* Patients with 300um ≤ the thickness of retina by optical coherence tomography
* Patients with visual acuity test ≥0.4 (20/50)
* Non-proliferative (background) retinopathy assessed by fundus photography and fluorescein angiography according to Airlie House Classification and ETDRS
* Patients with non-proliferative (background) retinopathy attested by the presence of Hard exudates within grade 2 and 5
* Patients with at leat one of the following lesions: Vascular leakages, Microaneurysms, Haemorrhages, Intraretinal microvascular abnormalities (IRMA)
* Patients with controlled Arterial Blood Pressure since the last 6 months (Diastolic Blood Pressure ≤90mmHg and Systolic Blood Pressure ≤130 mmHg) with or without medication
* Patients capable of conforming to the study protocol
* Patients who have given their free and informed consent
* The ability and willingness to comply with all study procedures

Exclusion Criteria:

* Diabetic Retinopathy which is being treated with laser therapy or should be treated with laser therapy before the end of the study
* Concomitant retinal disease due to causes other than diabetic microangiopathy
* Concomitant antihypertensive treatment, unless administered at stable dosage at least 6 months before the start of the study
* Concomitant Angiotensin-converting enzyme inhibitor / Angiotensin II receptor blocker therapy, unless administered at stable dosage for at least 6 months prior to the start of the study
* Concomitant Warfarin therapy
* Patients with laser therapy or intravitreal injection(avastin,steroid) within 3 months from enrolment
* Concomitant treatment with hemorrheological, vasoactive drugs and antithrombotics except acetylsalicylic acid at stable dosage
* Patients with severe liver impairment (Child-Pugh classification C)
* Patients with severe renal insufficiency (creatinine >2.2 mg/dl)
* Patients with severe cardiac insufficiency (New York Heart Association classes 3 - 4)
* Patients with clinical history of diathesis and haemorrhagic disease
* Individual hypersensitivity toward the product, heparin, low molecular weight heparin or heparin-like products
* Intended or ascertained pregnancy or lactation
* Participation to a trial within the past 6 months
* Surgery or trauma within the past 6 months
* Planned surgical intervention within 6 months from enrolment
* Patients unable to conform to the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2009-02; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Hard exudates | T12: 360 +/- 7 days from T0
  The lesion will be evaluated by fundus photography and fluorescein angiography, graded according to Modefied Airlie House Classification and ETDRS.

SECONDARY OUTCOMES:
microaneurysms | T12: 360 +/- 7 days from T0
  The lesion will be evaluated by fundus photography and fluorescein angiography, graded according to Modefied Airlie House Classification and ETDRS.
Vascular leakage | T12: 360 +/- 7 days from T0
  The lesion will be evaluated by fundus photography and fluorescein angiography, graded according to Modefied Airlie House Classification and ETDRS.
Haemorrhages | T12: 360 +/- 7 days from T0
  The lesion will be evaluated by fundus photography and fluorescein angiography, graded according to Modefied Airlie House Classification and ETDRS.
Intraretinal microvascular abnormalities (IRMA) | T12: 360 +/- 7 days from T0
  The lesion will be evaluated by fundus photography and fluorescein angiography, graded according to Modefied Airlie House Classification and ETDRS.

CONTACTS AND LOCATIONS:
Overall Officials: Ha Kyoung Kim, MD, Principal Investigator — Department of Ophthalmology, Kangnam Sacred Heart Hospital, College of Medicine, Hallym University
Locations (1):
- Kangnam Sacred Heart Hospital, Colloge of Medicine, Hallym University, Seoul, South Korea

REFERENCES:
- [Derived] Song JH, Chin HS, Kwon OW, Lim SJ, Kim HK; DRESS Research Group. Effect of sulodexide in patients with non-proliferative diabetic retinopathy: diabetic retinopathy sulodexide study (DRESS). Graefes Arch Clin Exp Ophthalmol. 2015 Jun;253(6):829-37. doi: 10.1007/s00417-014-2746-8. Epub 2014 Aug 12. PMID 25112845